CLINICAL TRIAL: NCT00126178
Title: A Multi-Center, Randomized, Phase 3 Study of Adjuvant Oncophage® Versus Observation in Patients With High Risk After Surgical Treatment for Renal Cell Carcinoma
Brief Title: Clinical Trial Studying a Personalized Cancer Vaccine in Patients With Non-metastatic Kidney Cancer
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: Agenus Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: C-100-12 Part 2
Record Dates: First submitted 2005-08-02; First posted 2005-08-03 (Estimated); Last update posted 2012-09-07 (Estimated); Status verified 2012-09

CONDITIONS: Kidney Cancer; Renal Cell Carcinoma
Keywords: Kidney Cancer; Renal; Immunotherapy; Vaccine
MeSH Terms: conditions — Kidney Neoplasms; Carcinoma, Renal Cell | interventions — vitespin

INTERVENTIONS:
Biological: HSPPC-96

SUMMARY:
This is an international, open label, randomized phase 3 trial in which patients with surgically removable kidney cancer will be randomly selected post-operatively to receive adjuvant treatment with autologous HSPPC-96 or no adjuvant treatment. All patients will undergo complete surgical removal of their tumors.

DETAILED DESCRIPTION:
This is an international, open label, randomized Phase 3 trial in which patients with surgically removable kidney cancer will be randomly selected post-operatively to receive adjuvant treatment with HSPPC-96 or no adjuvant treatment. All patients will undergo complete surgical removal of their tumors.

The primary objective of the study is to determine whether patients who receive adjuvant autologous HSPPC-96 (treatment group) after surgical resection of locally advanced renal cell carcinoma have improved recurrence-free survival as compared to patients who are not receiving adjuvant treatment (observation group). Eligible patients will have a 50% chance of receiving adjuvant treatment with HSPPC-96. Patients in the treatment arm of the trial will receive the vaccine once a week for 4 weeks, and then every other week until vaccine depletion or disease recurrence. Both groups of patients will be followed regularly for assessment of their disease status.

HSPPC-96 is an investigational, immunotherapeutic agent made from an individual patient's own tumor, which is collected at the time of surgery. A portion of the tumor tissue is sent to Antigenics' manufacturing facility where it will undergo processing to create a vaccine.

ELIGIBILITY:
This does not represent the full set of inclusion/exclusion criteria

Inclusion Criteria:

* Patients must have primary-intact resectable renal cell cancer, without distant metastasis and be scheduled to have surgery with curative intent
* Tumor size > 5 cm OR macroscopic nodes OR vena cava thrombus by radiologic evaluation
* At least 18 years old
* Signed informed consent

Exclusion Criteria:

* Prior surgery, chemo-, hormonal-, immuno-, or radiotherapy for kidney cancer
* History of other cancers within the last five years, with the exception of adequately treated cone-biopsied in situ carcinoma of the cervix uteri, basal or squamous cell carcinoma of the skin
* Current malignancies of any type in other sites
* No active uncontrolled infection, other serious medical illnesses, or splenectomy
* History of primary or secondary immunodeficiencies

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600
Dates: Start 2005-05; Primary Completion 2006-03 (Actual); Study Completion 2006-03 (Actual)

PRIMARY OUTCOMES:
To determine whether patients randomized to receive adjuvant HSPPC-96 (treatment) after surgical resection of the kidney cancer have improved recurrence-free survival as compared to patients who did not receive adjuvant treatment (observation)

SECONDARY OUTCOMES:
To determine whether patients randomized to receive adjuvant HSPPC-96 have improved overall survival as compared to patients in the observation group (without adjuvant treatment)
To further characterize the safety profile of HSPPC-96

CONTACTS AND LOCATIONS:
Locations (7):
- United States (5):
  - San Francisco, California
  - Stanford, California
  - Hackensack, New Jersey
  - San Antonio, Texas
  - South Burlington, Vermont
- Canada (2):
  - Victoria, British Columbia
  - Toronto, Ontario